CLINICAL TRIAL: NCT06493825
Title: Effects of Immersive Virtual Reality Mindfulness Application on Quality of Life, Anxiety and Depression Symptoms in Children With Severe Tinnitus and Misophonia - A Pilot Study
Brief Title: Mindfulness Application Effects on Mental Health Symptoms in Children With Severe Tinnitus and Misophonia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-0389
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Tinnitus; Misophonia
MeSH Terms: conditions — Tinnitus; misophonia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Subjects will undergo 4 weeks of immersive virtual reality exposure using the Aurora Mindfulness app (Invincikids) delivered using a Meta Quest 2 headset at the frequency of 10 minutes per session, 5 days out of a 7-day week. Subjects will undergo baseline, 2-week and 4-week measurement of symptoms using 5 validated instruments.
  Interventions: Other: Aurora Mindfulness app versus sham
- Placebo (Sham Comparator): Subjects will undergo 2 weeks of immersive virtual reality exposure using the Aurora Mindfulness sham app (Invincikids) delivered using a Meta Quest 2 headset at the frequency of 10 minutes per session, 5 days out of a 7-day week. Subjects will undergo baseline and 2-week measurement of symptoms using 5 validated instruments.
  Interventions: Other: Aurora Mindfulness app versus sham

INTERVENTIONS:
Other: Aurora Mindfulness app versus sham — It would either immersive virtual reality exposure for the experimental group or non-immersive virtual reality exposure for the placebo group.

SUMMARY:
Children with "bothersome" tinnitus and misophonia have elevated anxiety and depression symptoms. The mainstay therapy for adults and children with these disorders is cognitive behavioral therapy (CBT). CBT resources are expensive and scarce for the pediatric population. Immersive virtual reality (IVR) has been shown in the adult population to be a proxy for CBT for several mental health disorders. There is sufficient published evidence that IVR is useful in treating adults with anxiety and depression disorders. However, the evidence in children in treating either anxiety and depression symptoms or disorder is scant. Our group views IVR application as a promising medical device to decrease anxiety and depression scores in children with tinnitus and misophonia disorders.

This is a randomized placebo control (single-blinded to the study subjects) study in which there will be a 2:1 ratio between the experimental and placebo subjects, receiving either active IVR or placebo exposure. A total of 30 subjects with 20 experimental (10 tinnitus, 10 misophonia subjects) and 10 placebo (5 tinnitus and 5 misophonia subjects) will enroll in this randomized clinical trial. Assessment of change of quality of life, anxiety and depression symptoms will be based on 5 validated instruments.

The 5 validated instruments are: Tinnitus Functional Index (TFI), Amsterdam Misophonia Scale (A-MIS-S), Pediatric Quality of Life PEDQL), Screen for Child Anxiety Related Emotional Disorders (SCARED) and Short Mood and Feelings Questionnaire (SMFQ).

DETAILED DESCRIPTION:
Children with "bothersome" tinnitus and misophonia have elevated anxiety and depression symptoms. The mainstay therapy for adults and children with these disorders is cognitive behavioral therapy (CBT). CBT resources are expensive and scarce for the pediatric population. Immersive virtual reality (IVR) has been shown in the adult population to be a proxy for CBT for several mental health disorders. There is sufficient published evidence that IVR is useful in treating adults with anxiety and depression disorders. However, the evidence in children in treating either anxiety and depression symptoms or disorder is scant. Our group views IVR application as a promising medical device to decrease anxiety and depression scores in children with tinnitus and misophonia disorders.

This is a randomized placebo control (single-blinded to the study subjects) study in which there will be a 2:1 ratio between the experimental and placebo subjects, receiving either active IVR or placebo exposure. A total of 30 subjects with 20 experimental (10 tinnitus, 10 misophonia subjects) and 10 placebo (5 tinnitus and 5 misophonia subjects) will enroll in this randomized clinical trial. Assessment of change of quality of life, anxiety and depression symptoms will be based on 5 validated instruments.

The 5 validated instruments are: Tinnitus Functional Index (TFI), Amsterdam Misophonia Scale (A-MIS-S), Pediatric Quality of Life PEDQL), Screen for Child Anxiety Related Emotional Disorders (SCARED) and Short Mood and Feelings Questionnaire (SMFQ).

The primary outcome measures are the changes ot the pre-entry and post-entry scores of the 5 validated instruments at 2 weeks post-entry. In the experimental group, dose response will be measured between the 2- and 4-week results.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 10 to 18 years
* All genders and ethnicities
* Patients who meet criteria for "severe" symptoms of tinnitus and misophonia as scored by TIF and A-MISO-S

Exclusion Criteria:

* Severe developmental delay as not to understand verbal instructions necessary to complete the VR application/sham exposure.
* Severe visual impairment (refractive disorders are acceptable)
* Patients with unilateral or bilateral hearing loss of any type.
* History of seizure disorder

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Tinnitus Functional Index (TFI) | 2 weeks
  TFI measures the severity of tinnitus symptoms across several domains with a score range 0 to 90. The higher the score, the more dysfunction a subject is affected by tinnitus.
Amsterdam Misophonia Scale (A-MIS-S) | 2 weeks
  A-MIS-S measures the severity of misophonia symptoms across several domains with a score range of 0-24. The higher the score, the more dysfunction a subject is affected by misophonia.
Pediatric Quality of Life PedQL) | 2 weeks
  PedQL measures health-related quality of life of children with a range of 0 -100. The higher the score, the worse the health-related quality of life is.
Screen for Child Anxiety Related Emotional Disorders (SCARED) | 2 weeks
  SCARED screens for anxiety disorder in children and it ranges from 0-82. The higher the score, the higher the likelihood a child might have an anxiety disorder.
Short Mood and Feelings Questionnaire (SMFQ) | 2 weeks
  SMFQ measures depressive symptoms in children with a range of 0-26. The higher the score, the more depressive symptoms a child has.
Tinnitus Functional Index (TFI) | 4 weeka
  TFI measures the severity of tinnitus symptoms across several domains with a score range 0 to 90. The higher the score, the more dysfunction a subject is affected by tinnitus.
Amsterdam Misophonia Scale (A-MIS-S) | 4 weeks
  A-MIS-S measures the severity of misophonia symptoms across several domains with a score range of 0-24. The higher the score, the more dysfunction a subject is affected by misophonia.
Pediatric Quality of Life PedQL) | 4 weeks
  PedQL measures health-related quality of life of children with a range of 0 -100. The higher the score, the worse the health-related quality of life is.
Screen for Child Anxiety Related Emotional Disorders (SCARED) | 4 weeks
  SCARED screens for anxiety disorder in children and it ranges from 0-82. The higher the score, the higher the likelihood a child might have an anxiety disorder.
Short Mood and Feelings Questionnaire (SMFQ) | 4 weeks
  SMFQ measures depressive symptoms in children with a range of 0-26. The higher the score, the more depressive symptoms a child has.

SECONDARY OUTCOMES:
Satisfaction, acceptability and feasibility survey | 2 weeks
  The survey is in a 5-point Likert scale format with a range of very satisfied, satisfied, neutral, unsatisfied and very unsatisfied.
Satisfaction, acceptability and feasibility survey | 4 weeks
  The survey is in a 5-point Likert scale format with a range of very satisfied, satisfied, neutral, unsatisfied and very unsatisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No